CLINICAL TRIAL: NCT04702464
Title: A Phase 1, Open-label Study to Evaluate the Effect of a Dual CYP2C19 and CYP3A4 Inhibitor, Fluconazole, on the Pharmacokinetics of Fedratinib in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Effect of a Dual CYP2C19 and CYP3A4 Inhibitor, Fluconazole, on the Pharmacokinetics of Fedratinib in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: Impact Biomedicines, Inc., a wholly owned subsidiary of Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FEDR-CP-004; U1111-1261-2721 (Registry Identifier: WHO)
Expanded Access: NCT03723148 (Available)
Record Dates: First submitted 2020-12-23; First posted 2021-01-11 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Healthy Volunteers
Keywords: Healthy adult subjects; Fedratinib; CYP2C19; CYP3A4
MeSH Terms: interventions — fedratinib; Fluconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Administration (Experimental): * Day 1: Single dose of 100 mg fedratinib
  * Days 10 to 23, inclusive: Single dose of 400 mg fluconazole on Day 10 and once daily (QD) doses of 200 mg fluconazole on Days 11 to 23, inclusive
  * Day 18: Single dose of 100 mg fedratinib coadministered with the 200-mg fluconazole dose.
  Interventions: Drug: Fedratinib; Drug: Fluconazole

INTERVENTIONS:
Drug: Fedratinib — Fedratinib
Drug: Fluconazole — Fluconazole

SUMMARY:
This study is designed to test the effect of fluconazole (a dual CYP2C19 and CYP3A4 inhibitor) on the Pharmacokinetics (PK) of fedratinib. Knowledge of these effects can be used to determine if dose adjustments should be considered when fedratinib is coadministered with drugs that are dual CYP2C19 and CYP3A4 inhibitors.

Subjects will be screened for eligibility. Subjects who meet all inclusion criteria and none of the exclusion criteria will return to the clinical site on Day -1 for protocol-specified assessments, and will be domiciled at the clinical site from Day -1 to Day 27.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject must understand and voluntarily sign an informed consent form (ICF) prior to any study-related assessments/procedures being conducted.
2. Subject must be willing and able to communicate with the Investigator and adhere to the study visit schedule and other protocol requirements.
3. Subject is male or female of any race ≥ 18 to ≤ 65 years of age at the time of signing the ICF.
4. Female subjects NOT of childbearing potential must:

   a. Have been surgically sterilized (hysterectomy or bilateral oophorectomy; proper documentation required) at least 6 months before Screening, or postmenopausal (defined as 24 consecutive months without menses before Screening, with a follicle-stimulating hormone [FSH] level in the post-menopausal range according to the laboratory used at Screening).
5. Females of childbearing potential (FCBP1) must:

   1. Have a negative pregnancy test as verified by the investigator at Screening and Baseline (prior to starting study treatment). She must agree to ongoing pregnancy testing during the course of the study and after end of study treatment. This applies even if the subject practices true abstinence2 from heterosexual contact.
   2. Either commit to true abstinence from heterosexual contact (which must be reviewed on a monthly basis, as applicable, and source documented) or agree to use, and be able to comply with, any one of the following highly effective contraception methods without interruption, beginning at least 14 days prior to starting investigational product (IP), during the study treatment, and for at least 30 days after the last dose of IP.

      * Intrauterine device (IUD; non-hormonal only); tubal ligation; or a partner with a vasectomy. The chosen form of birth control must be effective by the time the subject receives the first dose of IP.
6. Male subjects must:

   a. Practice true abstinence from heterosexual contact (which must be reviewed on a monthly basis, as applicable, and source documented) or agree to use a barrier method of birth control (condoms not made from natural [animal] membrane [latex condoms are recommended]) during sexual contact with a pregnant female or FCBP while receiving study treatment, and for at least 30 days after the last dose of IP, even if he has undergone a successful vasectomy.
7. Must have a body mass index (BMI) ≥ 18 and ≤ 33 kg/m2 at screening.
8. Must be healthy, as determined by the Investigator on the basis of medical history, physical examination (PE), clinical laboratory test results, vital signs, and 12-lead electrocardiogram (ECG) at screening and check-in (Day -1), as applicable:

   Aspartate aminotransferase (AST), ALT, and total bilirubin must be at or below the upper limit of the reference range on or before check-in (Day -1). Other clinical laboratory results must be either within normal range or deemed not clinically significant by the Investigator. Any out of range lab tests may be repeated up to 1 time during Screening and up to 1 time at check-in per Investigator discretion to confirm eligibility.
9. Must be afebrile (febrile is defined as ≥ 38°C or 100.3°F).
10. Supine systolic blood pressure (BP) must be in the range of 90 to 150 mmHg (inclusive), supine diastolic BP must be in the range of 50 to 90 mmHg (inclusive), and pulse rate must be in the range of 45 to 90 bpm (inclusive) at Screening. Any out of range vital sign measurements may be repeated up to 1 time during Screening and up to 1 time at check-in per Investigator discretion to confirm eligibility.
11. Subject has a normal or clinically acceptable 12-lead ECG at screening; male subjects must have a corrected QT interval using Fridericia's formula (QTcF) value ≤ 430 msec and females must have a QTcF value ≤ 450 msec. An ECG may be repeated up to 2 times, and the average of the QTcF values will be used to determine subject eligibility.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. History (within 3 years prior to Screening) of any clinically significant neurological, GI, hepatic, renal, respiratory, cardiovascular, metabolic, endocrine, hematological, dermatological, psychological, or other major disorders as determined by the Investigator.
2. Any condition, including the presence of laboratory abnormalities, that places the subject at unacceptable risk if he or she were to participate in the study or confounds the ability to interpret data from the study (congenital nonhemolytic hyperbilirubinemia [eg, Gilbert's syndrome] is not acceptable).
3. Subject has prior history of Wernicke's Encephalopathy (WE).
4. Subject has signs or symptoms of WE (eg, ataxia, ocular paralysis, or cerebellar signs) without documented exclusion of WE by thiamine level and brain magnetic resonance imaging (MRI).
5. Subject has thiamine deficiency, defined as thiamine levels in whole blood below normal range according to institutional standard.
6. Use of any prescribed systemic or topical medication, including vaccines, within 30 days of the first dose administration (with the exception of ondansetron administered for purposes of this study).
7. Use of any nonprescribed systemic or topical medication (including vitamin/mineral supplements and herbal medicines) within 14 days of the first dose administration (with the exception of acetaminophen up to 2 grams/day for no more than 3 consecutive days to treat minor illness or headache [per Investigator judgment]).
8. Use of any metabolic enzyme or relevant transporter inhibitors or inducers that would affect the relevant drugs within 30 days of the first dose administration unless determined by the Investigator that there will be no impact on the study integrity or subject safety.

   The Indiana University "P450 Drug Interaction Table" should be used to determine inhibitors and/or inducers of metabolic enzymes (http://medicine.iupui.edu/clinpharm/ddis/table/aspx). The Sponsor should be contacted for questions about potential drug-drug interactions and exclusions/prohibitions when necessary.
9. Exposure to an investigational drug (new chemical entity) within 30 days preceding the first dose administration or 5 half-lives of that investigational drug, if known (whichever is longer).
10. Presence of any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism, and excretion (eg, bariatric procedure, cholecystectomy). Appendectomy is acceptable.
11. Donated blood or plasma within 8 weeks before the first dose administration.
12. History of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual [DSM]) within 2 years before dosing or positive drug screening test reflecting consumption of illicit drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2021-05-09 (Actual); Study Completion 2021-05-13 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic - Maximum observed plasma concentration (Cmax) for Fedratinib | Up to 216 hours following the last dose of fedratinib
  Maximum observed plasma concentration
Pharmacokinetic - Area under the plasma concentration-time curve (AUC) for Fedratinib | Up to 216 hours following the last dose of fedratinib
  Area under the plasma concentration-time curve

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | From enrollment until at least 30 days after completion of study treatment
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a pre-existing condition) should be considered an AE.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PPD Phase 1 Clinic, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/

REFERENCES:
- [Derived] Chen Y, Ogasawara K, Wood-Horrall R, Thomas M, Thomas M, He B, Liu L, Xue Y, Surapaneni S, Carayannopoulos LN, Zhou S, Palmisano M, Krishna G. Effect of fluconazole on the pharmacokinetics of a single dose of fedratinib in healthy adults. Cancer Chemother Pharmacol. 2022 Oct;90(4):325-334. doi: 10.1007/s00280-022-04464-w. Epub 2022 Aug 24. PMID 36001108